CLINICAL TRIAL: NCT05924490
Title: Cognitive Engagement and Aging Mind: A Randomized Control Trial to Determine the Effects of Adaptive Real-time Strategy Game Training on Cognition and Brain Functions of Older Adults
Brief Title: Cognitive Engagement and Aging Mind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 12-57
Record Dates: First submitted 2021-05-07; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2021-05

CONDITIONS: Age-related Cognitive Decline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time strategy-based videogame training (Experimental): Participants played a real-time strategy-based videogame in laboratory setting, Rise of Nations, for 2 hours a day, two days per week, for 5 weeks.
  Interventions: Behavioral: Real-time strategy-based videogame training
- Crystallized intelligence training (Active Comparator): Participants completed a series of crossword puzzles each week, for 5-6 weeks. Training sessions were completed at the participants' home or area of preference. Participant received a periodic phone call (2 times per week) from research staff to update any notes or details regarding participants' study progress.
  Interventions: Behavioral: Semantic Knowledge training

INTERVENTIONS:
Behavioral: Real-time strategy-based videogame training — Rise of Nation is a complex strategy-based video game, in which individualized-adaptive feedbacks are constantly given to players based on their performance.
  Arms: Real-time strategy-based videogame training
Behavioral: Semantic Knowledge training — Packages of various cross-word puzzles include word search, word ladder, and word wheel.
  Arms: Crystallized intelligence training

SUMMARY:
The purpose of this research is to examine whether and to what extent training of different types of cognitive engagement will improve performance on fluid cognitive abilities that typically decline with age. The research covered by this protocol will use behavioral data that yield response latencies and accuracies of the untrained tasks, and brain activations in fMRI tasks, to test specific hypotheses about neural plasticity and cognitive plasticity from these engagement techniques. Hence, human subjects will be employed in an experiment lasting for 20 hours spanning over 2 months where they will either receive real-time strategy-based videogame training or crystallized intelligence training. In addition, long-term retention data will be obtained after 6 month post-training to investigate any long-term benefits.

DETAILED DESCRIPTION:
The purpose of this research is to examine whether and to what extent training of different types of cognitive engagement will improve performance on fluid cognitive abilities that typically decline with age (such as, speed of information processing, working memory capacity, episodic memory, and executive functions). The research covered by this protocol will use behavioral data that yield response latencies and accuracies of the untrained tasks, and brain activations in fMRI tasks, to test specific hypotheses about the extent of transfer, if any, and the underlying cognitive constructs that may be trained in the process. Hence, human subjects will be employed in an experiment lasting for 20 hours spanning over 2 months where they will either receive real-time strategy-based videogame training or crystallized intelligence training. In addition, long-term retention data will be obtained after 6 month post-training to investigate any long-term benefits.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* over 50 Years of Age
* native or fluent English speaker
* not Color-blind
* Magnetic Resonance Imaging eligible
* Mini Mental Status Examination Score >24

Exclusion Criteria:

* Left-handed or ambidextrous
* younger than 50
* cannot distinguish colors during color blindness test
* claustrophobia
* metal artifact in body
* over 300 lb
* pacemaker
* MMSE score lower than 24
* history of stroke
* history of substance or alcohol abuse
* currently taking anti-psychotic or anti-depression medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Immediate change in the composite score of executive functions | 9-11 weeks
  Change in the composite score of executive functions, and its subcomponents, from baseline to post-training. Higher change in score represents better outcome.
Immediate change in the composite score of episodic memory | 9-11 weeks
  Change in the composite score of episodic memory from baseline to post-training.Higher change in score represents better outcome.
Immediate change in brain activations during executive functions: multi-tasking | 9-11 weeks
  Change in fMRI brain activations from baseline to post-training.
Immediate change in brain activations during executive functions: working memory updating | 9-11 weeks
  Change in fMRI brain activations from baseline to post-training.

SECONDARY OUTCOMES:
Immediate change in the composite score of working memory capacity | 9-11 weeks
  Change in the composite score of working memory capacity from baseline to post-training.Higher change in score represents better outcome.
Immediate change in the fluid reasoning measure | 9-11 weeks
  Change in the fluid reasoning measure (Raven's Advanced Progressive Matrices, a paper and pencil test) from baseline to post-training. Higher change in score represents better outcome.
immediate change in the composite score of cognition | 9-11 weeks
  Change in composite score of cognition from baseline to long-term retention. Composite score for overall cognition is summed across composite scores for executive function, processing speed, processing speed, working memory capacity and fluid reasoning. Higher change in score represents better outcome.

OTHER OUTCOMES:
Immediate change in the processing speed construct | 9-11 weeks
  Change in the processing speed construct from baseline to post-training. Higher change in score represents better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chandramallika Basak, Ph.D., Principal Investigator — The University of Texas at Dallas
Locations (1):
- The Center for Vital Longevity (UT Dallas), Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is not a federally funded data, so no IDP is planned to be shared. However, all descriptive statistics will be provided in the publications, therefore, all meaningful data for the outcomes will be reported for any future meta-analyses or calculations of effect size.